CLINICAL TRIAL: NCT03232879
Title: Combining Motor Imagery With Action Observation Does Not Lead to a Greater Autonomic Response Than Motor Imagery Alone During Simple and Functional Movements: a Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Autonomic Nervous System
Keywords: Motor Imagery; Action Observation; Heart Rate; Respiration Rate; Electrodermal Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental 1 (Experimental): Motor Imagery
  Interventions: Behavioral: Motor Imagery
- Experimental 2 (Experimental): Action Observation
  Interventions: Behavioral: Action Observation
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Motor Imagery — Two consecutive 30 seconds imagery tasks were performed, both based on two movements that are recorded in the Revised Movement Imagery Questionnaire (MIQ-R).
  Arms: Experimental 1
Behavioral: Action Observation — Two consecutive 30 seconds imagery tasks were performed, both based on two movements that are recorded in the Revised Movement Imagery Questionnaire (MIQ-R). Before the subjects performed the mental MI practice, they were presented with a 30 seconds video that displayed the task that they ought to imagine later. A video was played prior to the first practice of imagination and after the second mental practice, a second video was shown.
  Arms: Experimental 2

SUMMARY:
The main objective of this study was to compare the activation of the Sympathetic Nervous System in a program that combined Motor Imagery with Action Observation, in contrast to an isolated Motor Imagery program on the one hand in asymptomatic subjects and in the other hand in patients with chronic low back pain.

DETAILED DESCRIPTION:
Motor Imagery (MI) is defined as a dynamic mental process that involves the representation of an action, in an internal way, without its actual motor execution. The Action Observation (AO) evokes an internal, real-time motor simulation of the movements that the observer is perceiving visually. Both mental processes trigger the activation of the neurocognitive mechanisms that underlie the planning and execution of voluntary movements in a manner that resembles how the action is performed in a real manner.

Both observation and imagination share a great number of common mental processes based primarily on sensory perception, and the information stored by memory systems. The activation of the motor command during a mental practice does not induce an active movement probably due to an inhibitory mechanism in the primary motor cortex on the descending corticospinal tract pathways. However, this inhibition is not complete, for it is well known that the training of mental practice involves a component of the autonomic nervous system (ANS).

It has been shown that both MI and AO lead to changes in the ANS that cause excitatory sympathetic responses, although the neurophysiological bases remain uncertain and are still based on hypotheses. The functional relations between both neurocognitive processes and the sympathetic-excitatory nervous system (SNS) could be based on a preparation phase in which, the activation of the SNS, happens to a near effort and, therefore, to a close energy expenditure in physiological processes (i.e., cardiorespiratory adaptationse) which will take place in order to face said metabolic changes produced by the voluntary movement itself. In addition, several hypotheses have been described regarding the notion that the SNS not only has the quantitative objective of providing energy to the muscle effectors, but that it also qualitatively and specifically designs and adapts the parameters on demand in an attempt to save the energy provided for each precise motor execution.

Taking into account that both MI and AO cause sympathetic-excitatory changes that induce an increase in heart rate, blood pressure, respiratory rate, electrodermal activity , our hypothesis is that the combination of MI and AO induces an autonomic sympathetic-excitatory shift greater than MI does in isolation. Therefore, the main objective of this study was to compare the results obtained from intervention groups on the subject of the activation of the SNS in a program that combined MI with AO, in contrast to an isolated MI program on the one hand in asymptomatic subjects and in the other hand in patients with chronic low back pain.. The secondary objective of the present study was to explore whether there is any relationship between the sympathetic-excitatory response and the ability to generate motor imagery, the mental chronometry, and the level of physical activity.

ELIGIBILITY:
Inclusion Criteria asymptomatic subjects:

* Age between 18 and 60
* Healthy and with no pain subjects

Inclusion Criteria patients with chronic low back pain:

* Low back pain for at least the prior 3 months
* Low back pain of nonspecific nature
* Age between 18 and 60
* Low back pain for at least 10 days per month
* Intensity of pain of between 3 and 10 on the Visual Analogue Scale

Exclusion Criteria asymptomatic subjects:

* Any cognitive impairment that hindered viewing of audiovisual material.
* Difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.
* Underage subjects
* Subjects with pain at the time of the study.

Exclusion Criteria patients with chronic low back pain:

* Any cognitive impairment that hindered viewing of audiovisual material.
* Difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.
* Underage subjects
* Having undergone back surgery
* Specific spinal pathology
* Recent trauma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Electrodermal Activity | Change in electrodermal activity after 5 minutes post-intervention
  Electrodermal Activity will be measured through the use of two electrodes that recorded changes in conductance through the skin located at the back of the dominant hand
Respiration Rate | Change in respiration rate after 5 minutes post-intervention
  Respiration Rate will be measured through a pressure transducer located in the centre of the chest, where it was fixed by a strap
Heart Rate | Change in heart rate after 5 minutes post-intervention
  Heart Rate will be measured by three electrodes located in the left area of the chest. One of the electrodes was placed in the middle zone while a second electrode was positioned on the lateral side, and a third one on the lower left side, below the first electrode.

SECONDARY OUTCOMES:
Visual and Kinesthetic Motor Imagery Ability | Pre-intervention
  Visual and Kinesthetic Motor Imagery Ability will be measured with MIQ-R Questionnaire. MIQ-R has 4 movements repeated in two subscales, a visual and a kinaesthetic one. Additionally, a score between 1 and 7 is assigned, with 1 representing difficulty in picturing the motor image or difficulty in feeling the movement previously made, and 7 representing the maximum ease. A modification was made in the MIQ-R. Items 2 and 5, in which a small jump is made, were changed by standing on tiptoe. The internal consistencies of the MIQ-R have been consistently adequate with Cronbach's α coefficients ranging above 0.84 for the total scale, 0.80 for de visual subscale and 0.84 for the kinesthetic subscale.
Mental Chronometry | Pre-intervention
  Mental chronometry evaluation was also used to measure the subject's motor imagery ability. Using a stopwatch, the time spent for performing each MIQ-R task was recorded. Time recorded corresponds to the interval between the command to start the task, given by the evaluator, and the verbal response of conclusion of the task, given by the subject. Mental chronometry is a reliable behavioral task that has previously been employed to collect an objective measure of MI ability
The degree of physical activity | Pre-intervention
  The degree of physical activity was objectified through the The International Physical Activity Questionnaire questionnaire, which allows the subjects to be divided into three groups according to their level of activity, which can be high, moderate, and low or inactive

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No